CLINICAL TRIAL: NCT05441176
Title: TULIP et MASC : Premiers Usages
Acronym: TEMPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A01451-42
Record Dates: First submitted 2022-06-23; First posted 2022-07-01 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Thoracic Outlet Syndrome
Keywords: suspicion of arterial TOS and/or veinous TOS; DASH questionnaire; TULIP and MASC questionnaires
MeSH Terms: conditions — Thoracic Outlet Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with suspicion of TOS (Experimental): Patients coming for a visit to diagnostic TOS and submitted TULIP and MASC questionnaires
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Scoring of the DASH is performed according to references.

SUMMARY:
The aim of this work is to propose two new questionnaires (TULIP and MASC) which are simple to complete by the patient, quick to analyze and can be calculated directly by the physician, adapted to the general population, whether during an initial evaluation or for follow-up.

The TULIP questionnaire aims to characterize the symptoms suggestive of Thoracic Outlet Syndrome (TOS). The MASC questionnaire aims to assess the functional maintenance of TOS in a simpler way (fewer questions) than the Disability of the Arm, Shoulder and Hand (DASH) questionnaire and in a lateralized way.

DETAILED DESCRIPTION:
Two questionnaires the TULIP and the MASC are submitted (self completion) to patients suspected of TOS.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of Thoracic Outlet Syndrome

Exclusion Criteria:

Non applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of both questionnaires : percentage of questionnaires correctly completed | 1 day
  Estimation of the percentage of questionnaires correctly completed. "correctly completed" means a questionnaire without physician's correction.

SECONDARY OUTCOMES:
TULIP : Diagnostic performance of vascular TOS by concordance between each response and vascular investigations results evaluation | 1 day
  Determine the diagnostic performance of each response according to the presence or absence of vascular compression of the arm considered.
  We evaluate the correlation between each response of TULIP's items and vascular investigation results (positive ultrasound or/and angiography)
MASC : Concording with DASH questionnaire | 1 day
  Correlation coefficient with the DASH questionnaire
MASC : Comparison between concordance MASC/DASH and concordance MASC/Quick DASH | 1 day
  Comparison of correlation coefficient with the DASH questionnaire and of correlation coefficient with the Quick-DASH questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Angers, France